CLINICAL TRIAL: NCT05492357
Title: The Effect of Recurrent Application of Liquid Platelet-rich Fibrin in the Extraction Socket on the Hard and Soft Tissues. A Randomised Controlled Trial
Brief Title: Effects of Recurrent Application of Liquid-PRF on Hard and Soft Tissues
Acronym: Liquid-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cezar Edward Lahham (Other)
Responsible Party: Sponsor-Investigator, Cezar Edward Lahham, Principal Investigator, Arab American University (Palestine)
Organization: Arab American University (Palestine) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC/HC/1151/22
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Liquid-PRF; A-PRF Plus
Keywords: recurrent; Liquid platelet-rich fibrin; Advanced platelet-rich fibrin plus; ridge preservation
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Human patients:
  20 patients who need tooth/ teeth extraction would be selected according to the following criteria:
  INCLUSION CRITERIA:
  1. Men and women over 18 years of age
  2. Indication of a simple extraction
  3. Delivery of signed informed consent
  EXCLUSION CRITERIA:
  1. Need for multiple extractions
  2. Presence of severe swelling prior to surgery in the extraction area
  3. Regular treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or other anti-inflammatory drugs
  4. Presence of hematologic disease
  5. Previous radiation, chemotherapy, or immunosuppressive treatments
  6. Uncontrolled diabetes mellitus, metabolic bone disease, ongoing treatment with bisphosphonates drugs, or pregnancy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Advanced platelet-rich fibrin plus + Liquid platelet-rich fibrin (Experimental): A-PRF plus + Liquid-PRF are prepared from the patient's blood.
  Interventions: Other: Liquid platelet-rich fibrin; Other: Advanced Platelet-rich fibrin plus
- Advanced platelet-rich fibrin plus alone (Experimental): A-PRF+ is prepared from the patient's blood.
  Interventions: Other: Advanced Platelet-rich fibrin plus

INTERVENTIONS:
Other: Liquid platelet-rich fibrin — Liquid platelet-rich fibrin is prepared from the patient's blood and injected into the extraction socket every two weeks (up to 3 months = Just 4 times of application)
  Other Names: Liquid-PRF
  Arms: Advanced platelet-rich fibrin plus + Liquid platelet-rich fibrin
Other: Advanced Platelet-rich fibrin plus — A-PRF+ is placed into the extraction socket immediately after tooth extraction

SUMMARY:
Procedure: Tooth is extracted, then A-PRF+ is placed inside the socket. After that the ridge dimensions is asses clinically at the baseline) in addition to clinical assessment of the gingival biotype at the baseline.

Then patients will be divided into 2 groups:

Group 1: 50% of patients will have recurrent Liquid-PRF injections inside the extraction socket every 2 weeks (A-PRF+, followed by recurrent Liquid-PRF) Group 2: 50% of patients without recurrent (just A-PRF+) After 3 months from extraction: both groups will be assessed clinically (gingival biotype) & (Ridge dimensions) in order to assess the role of recurrent application of Liquid-PRF on these parameters.

DETAILED DESCRIPTION:
In this study, we will select 20 patients who need a simple tooth extraction, then determine the gingival biotype, take a blood sample to prepare A-PRF+ (centrifugation of the patient's blood for 8 min at 1300 rpm using red caps tubes), then do the extraction. After that, A-PRF+ is prepared and inserted into the extraction socket, and sutured using horizontal mattress suturing technique.

After the clinical assessment of the ridge dimensions at the baseline

Then patients will be divided into 2 groups:

Group 1: 10 patients will have recurrent Liquid-PRF injections inside the extraction socket every 2 weeks (A-PRF+, followed by recurrent Liquid-PRF) Liquid-PRF preparation: Centrifugation of the patient's blood for 8 min at 2500 rpm using white caps tubes.

Group 2: 10 patients without recurrent application of Liquid-PRF (just A-PRF+) After 3 months from extraction: both groups will be assessed clinically (gingival biotype) & (Ridge dimensions) in order to evaluate the effect of recurrent application of Liquid-PRF on these parameters.

Assessment method:

for Hard tissue evaluation (Bone): we assess the dimensions clinically For soft tissue: we will use a periodontal probe to assess the gingival thickness after giving local anesthesia.

---------------------------------------------

Selection Criteria

INCLUSION CRITERIA:

1. Men and women over 18 years of age
2. Indication of a simple extraction
3. Delivery of signed informed consent

EXCLUSION CRITERIA:

1. Need for multiple extractions
2. Presence of severe swelling prior to surgery in the extraction area
3. Regular treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or other anti-inflammatory drugs
4. Presence of hematologic disease
5. Previous radiation, chemotherapy, or immunosuppressive treatments
6. Uncontrolled diabetes mellitus, metabolic bone disease, ongoing treatment with bisphosphonates drugs, or pregnancy

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age
2. Indication of a simple extraction (Non-molar tooth)
3. Delivery of signed informed consent
4. Need delayed implant placement in the place of extraction

Exclusion Criteria:

1. Need for multiple extractions
2. Presence of severe swelling prior to surgery in the extraction area
3. Regular treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or other anti-inflammatory drugs
4. Presence of hematologic disease
5. Previous radiation, chemotherapy, or immunosuppressive treatments
6. Uncontrolled diabetes mellitus, metabolic bone disease, ongoing treatment with bisphosphonates drugs, or pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Ridge dimensions | 3 months
  assessment of ridge dimensions 3 months after intervention for both groups. At the baseline it was assessed clinically. After 3 months, the flap was released and the ridge width and height were assessed clinically.
Gingival biotype | 3 months
  assessment of gingival biotype 3 months after intervention according to gingival thickness (using periodontal probe: if <1 mm = Thin, while if >1 =Thick).

CONTACTS AND LOCATIONS:
Locations (1):
- Cezar Lahham, Bethlehem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lahham C, Ta'a MA, Lahham E, Michael S, Zarif W. The effect of recurrent application of concentrated platelet-rich fibrin inside the extraction socket on the hard and soft tissues. a randomized controlled trial. BMC Oral Health. 2023 Sep 19;23(1):677. doi: 10.1186/s12903-023-03400-5. PMID 37726689